CLINICAL TRIAL: NCT05604196
Title: Searching for Biomarkers of Metabolic Obesity.
Brief Title: Biomarkers of Metabolic Obesity.
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: SUB/3/DN/20/001/3316; SUB/3/DN/21/001/3316 (Other Grant/Funding Number: Medical University of Bialystok)
Record Dates: First submitted 2022-10-25; First posted 2022-11-03 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: obesity; saliva; blood serum; BMI; proinflammatory cytokines; proinflammatory adipokines; IL-6; IL-23; IL-1beta; resistin; TNF-alpha; MMP-2; MMP-9
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STUDY GROUP: Study group included 79 people (48 women and 31 men), with BMI = 30.0-39.9 kg / m2) and excessive total body fat percent (TBF%) content (>30% TBF women and >25% TBF men).
- CONTROL GROUP: Control group included 41 people (31 women and 10 men), with BMI = 18.5-24.9 kg / m2) and normal total body fat percent (TBF%) content (20-30% TBF women and 15-20% TBF men).

SUMMARY:
The main aims of the work: Analysis of the concentration of selected pro-inflammatory parameters in blood serum and saliva of people with different distribution of subcutaneous and visceral adipose tissue. Analysis of metabolic obesity biomarkers in saliva and blood serum. Evaluation of new diagnostic methods for the early determination of the risk of metabolic obesity and its complications.

Based on the inclusion and exclusion criteria the observational study was conducted among 119 people (79 women and 41 men). Study group included 79 people (48 women and 31 men with obesity), and control group included 41 people (31 women and 10 men with normal body weight).

The study consisted of three visits. The first included qualification for the study, body composition measurements, ankle-brachial index test and completing the questionnaires and 3-day nutrition diaries. At the second visit blood was collected to conduct the morphological test. At the third visit saliva was collected to determine the proinflammatory cytokine and adipokine concentration.

DETAILED DESCRIPTION:
The main aims of the work:

1. Analysis of the concentration of selected pro-inflammatory parameters in blood serum and saliva of people with different distribution of subcutaneous and visceral adipose tissue.
2. Analysis of metabolic obesity biomarkers in saliva and blood serum.
3. Evaluation of new diagnostic methods for the early determination of the risk of metabolic obesity and its complications.

The study protocol was approved by the Bioethics Committee of the Medical University, no. R-I-002/647/2019 and APK.002.39.2021. All participants gave informed written consent to participate in the study before its commencement. The study began in January 2020 and ended in May 2022.

The research was carried out at the Department of Dietetics and Clinical Nutrition (Faculty of Health Sciences of the Medical University of Bialystok), Biochemical Diagnostics Department (University Clinical Hospital in Bialystok), as well as at the Department of Biotechnology (Faculty of Pharmacy with the Division of Laboratory Medicine of the Medical University of Bialystok).

The first visit took place in the Department of Dietetics and Clinical Nutrition at the Medical University of Bialystok. It included qualification for the study based on the inclusion and exclusion criteria, discussion of the purpose of the study and signing the written consent for the study by the participants, as well as information about the protection of their personal data and full anonymity. 200 people volunteered for the study. Based on the inclusion and exclusion criteria the observational study was conducted among 119 people (79 women and 41 men). Each participant received an individual code (e.g. A01, A02, B01, B02 etc.), which was used to identify the participants in further stages of the study.

All participants completed: The World Health Organization Quality of Life (WHOQOL- BREF) survey, International Physical Activity Questionnaire - IPAQ, Beliefs and Eating Habits Questionnaire created by Behavioral Conditions of Nutrition Team, Committee of Human Nutrition Science, Polish Academy of Science, and 3-day Nutrition Diary (participants described meals consumed for the next three days, including two working days and one day off).

The participants of the study had measurements of anthropometric parameters (body weight, height, waist and hip circumference) and the BMI (Body Mass Index) was calculated. On its basis the participants were divided into the study and control group. Moreover, the WHR ratio (Waist to Hip Ratio), WHtR ratio (Waist to Height Ratio) and RFM ratio (Relative Fat Mass) were calculated.

In order to determine the body composition of the study participants, an electrical bioimpedance body composition analysis was carried out using the devices: BioScan 920-2 (Great Britain, Essex) and InBody 270 (South Korea, Seoul). The examination was performed in the morning, fasting, without any intense physical exertion.

An ankle-brachial index test (MESI, Cracow, Poland) compares the blood pressure measured at the ankle with the blood pressure measured at the arm was also used in the study. This analysis was performed to assess the risk of lower limb atherosclerosis. Moreover blood pressure and resting heart rate using an electric sphygmomanometer was measured for all the study participants.

The second visit took place at the Biochemical Diagnostics Department (University Clinical Hospital in Bialystok). 10 ml of venous blood were collected from all participants in the study. Oral glucose tolerance test (OGTT) was performed, and on its basis, the concentration of glucose and insulin was determined (fasting, and after 60 and 120 minutes of the test). Concentrations of total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride, C-reactive protein, glucose, insulin, serum urea, serum creatinine, serum uric acid, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) was assessed on ALINITY ci, Abbott.

Blood samples were taken patients and frozen at -80 °C. Serum levels of total adiponectin (Quantikine ELISA Human Total Adiponectin/Acrp30 Immunoassay, R&D Systems, Abingdon, UK), resistin (Quantikine ELISA Human Resistin Immunoassay, R&D Systems, Abingdon, UK), IL-6 (Quantikine ELISA Human IL-6 Immunoassay, R&D Systems, Abingdon, UK), TNFα (Quantikine ELISA Human TNFα Immunoassay, R&D Systems, Abingdon, UK), IL-1β (Quantikine ELISA Human IL-1β/IL-1F2 Immunoassay, R&D Systems, Abingdon, UK), IL-23 (Quantikine ELISA Human IL-23 Immunoassay, R&D Systems, Abingdon, UK), MMP-9 (Quantikine ELISA Human MMP-9 Immunoassay, R&D Systems, Abingdon, UK) and total MMP-2 (Quantikine ELISA Total MMP-2 Immunoassay, R&D Systems, Abingdon, UK) were assessed with the enzyme-linked immunosorbent assay (ELISA) according to the manufactures' instructions.

The third visit took place at the Department of Biotechnology (Faculty of Pharmacy with the Division of Laboratory Medicine of the Medical University of Bialystok).

Saliva was collected using a standard method. Samples from the subjects were collected between 9:00 and 11:00 a.m. All subjects abstained from eating and drinking for 2 h. The subjects rinsed their mouths with deionized water and were sitting in a comfortable position with their eyes open and head titled slightly forward. Unstimulated whole saliva was collected for 10 min by spitting described by Navazesh. Saliva samples were homogenized and clarified by centrifugation at 1200 RPMI for 15 min at 4°C. The aliquots of clarified supernatants were stored at -70 °C for the ELISA measurements.

Highly sensitive assay kits (R&D Systems, Minneapolis, USA) were used to determine the concentrations of IL-6, IL-1β, IL-23, resistin, MMP-9, MMP-2 and TNF-α in the salivary samples from the study participants. The tests were carried out according to the manufacturer's protocols. The microtiter plate provided in kits was pre-coated with monoclonal antibody specific for analyzed protein. Standards and samples were added to the appropriate microtiter plate wells. After the incubation at room temperature, enzyme-linked polyclonal antibody was added. Then, the microplate wells were aspirated and washed four times. Next, a substrate solution was added to each well. The enzyme-substrate reaction was terminated by the addition of a stop solution and the color change was measured spectrophotometrically at 450 nm ±2 nm. The antigen concentration in the samples was determined by comparing the O.D. to the standard curve. The antigen concentration in the samples was determined by comparing the O.D. to the standard curve.

ELIGIBILITY:
Inclusion Criteria:

* women and men aged 20-55
* primary obesity
* certificate from the dentist confirming the absence of periodontitis and inflammation in the oral cavity.

Exclusion Criteria:

* secondary obesity,
* type I and II diabetes,
* exacerbated coronary artery disease,
* endocrine disorders,
* eating disorders,
* pregnancy and lactation period,
* use of hormonal contraception or hormone replacement therapy, steroid therapy, antiretroviral therapy,
* surgical or pharmacological history obesity treatment,
* pacemaker

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 200 people volunteered for the study. The participants came from the Podlaskie Voivodeship, Poland. The first visit took place in the Department of Dietetics and Clinical Nutrition at the Medical University of Bialystok. Based on the inclusion and exclusion criteria the observational study was conducted among 119 people (79 women and 41 men).
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Analysis of the concentration of selected pro-inflammatory cytokines and adipokines in the saliva of patients with normal and excess body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  Analysis of the concentration in saliva of MMP-9, MMP-2, IL-6, TNF-α, resistin, IL-1β, IL-23 in patients with normal and excess body weight (obesity).
Analysis of the concentration of selected pro-inflammatory cytokines and adipokines in the blood serum of patients with normal and excess body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  Analysis of the concentration in saliva of adiponectin, IL-6,TNF-α, MMP-9, MMP-2, resistin, IL-1β, IL-23 in patients with normal and excess body weight (obesity).
Analysis of body composition of people with normal and excess body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  In order to determine the body composition of the study participants, an electrical bioimpedance body composition analysis was carried out using the InBody 270 (South Korea, Seoul) device, which enabled the assessment of the following parameters: total body fat percentage, total lean body mass percentage, total body fat mass, total skeletal muscle mass, total body water (L), extracellular (L) and intracellular (L) water.
Analysis of body composition and adipose tissue redistribution of people with normal and excess body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  In order to determine the body composition of the study participants an electrical bioimpedance body composition analysis was carried out using the device: BioScan 920-2 (Great Britain, Essex), which enabled the assessment of the following parameters: total body fat percentage, total lean body mass percentage, total body fat mass, total skeletal muscle mass, total body water (L), extracellular (L) and intracellular (L) water. Also, the area of adipose tissue in the abdominal cross-section was determined: visceral (VAT- Visceral Adipose Tissue) and subcutaneous (SAT- Subcutaneous Adipose Tissue), and visceral to subcutaneous fat ratio (VAT / SAT ratio).
Analysis of differences in the eating habits of people with normal and excessive body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  All participants completed "Beliefs and Eating Habits Questionnaire" created by Behavioral Conditions of Nutrition Team Committee of Human Nutrition Science, Polish Academy of Science.
Analysis of differences in the diet of people with normal and excessive body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  All participants completed 3-day Nutrition Diary.
Analysis of differences in physical activity of people with normal and excessive body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  All participants completed "International Physical Activity Questionnaire - IPAQ".
Analysis of differences in quality of life of people with normal and excessive body weight (obesity). | 24 months (analyzes were performed throughout the study period).
  All participants completed The World Health Organization Quality of Life (WHOQOL- BREF) survey.
Risk assessment of lower limb atherosclerosis. | 24 months (analyzes were performed throughout the study period).
  An ankle-brachial index test compares the blood pressure measured at the ankle with the blood pressure measured at the arm was used in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Ostrowska, Professor, Principal Investigator — Department of Dietetics and Clinical Nutrition Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Poland

REFERENCES:
- [Background] Zhang CZ, Cheng XQ, Li JY, Zhang P, Yi P, Xu X, Zhou XD. Saliva in the diagnosis of diseases. Int J Oral Sci. 2016 Sep 29;8(3):133-7. doi: 10.1038/ijos.2016.38. PMID 27585820
- [Background] Duffles LF, Hermont AP, Abreu LG, Pordeus IA, Silva TA. Association between obesity and adipokines levels in saliva and gingival crevicular fluid: A systematic review and meta-analysis. J Evid Based Med. 2019 Nov;12(4):313-324. doi: 10.1111/jebm.12363. Epub 2019 Sep 4. PMID 31482694
- [Background] Zysk B, Ostrowska L, Smarkusz-Zarzecka J. Salivary Adipokine and Cytokine Levels as Potential Markers for the Development of Obesity and Metabolic Disorders. Int J Mol Sci. 2021 Oct 28;22(21):11703. doi: 10.3390/ijms222111703. PMID 34769133
- [Background] Kunz HE, Hart CR, Gries KJ, Parvizi M, Laurenti M, Dalla Man C, Moore N, Zhang X, Ryan Z, Polley EC, Jensen MD, Vella A, Lanza IR. Adipose tissue macrophage populations and inflammation are associated with systemic inflammation and insulin resistance in obesity. Am J Physiol Endocrinol Metab. 2021 Jul 1;321(1):E105-E121. doi: 10.1152/ajpendo.00070.2021. Epub 2021 May 17. PMID 33998291
- [Background] Ostrowska L, Gornowicz A, Pietraszewska B, Bielawski K, Bielawska A. Which salivary components can differentiate metabolic obesity? PLoS One. 2020 Jun 29;15(6):e0235358. doi: 10.1371/journal.pone.0235358. eCollection 2020. PMID 32598403
- See also: World Health Assembly: Follow-up to the Political Declaration of the High-level Meeting of the General Assembly on the Prevention and Control of Non-communicable Diseases. (Paper WHA66.10) 2013, 1-55. — http://apps.who.int/gb/ebwha/pdf_files/WHA66/A66_R10-en.pdf
- See also: World Obesity Federation: Global trends in obesity. [in:] Obesity: missing the 2025 global targets. Trends, Costs and Country Reports 2020, 16-33. — http://www.worldobesity.org/resources/resource-library/world-obesity-day-missing-the-targets-report